CLINICAL TRIAL: NCT06423963
Title: Remote Exercise and Nutritional Prehabilitation for Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23088
Record Dates: First submitted 2024-04-22; First posted 2024-05-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity, nutrition counseling and monitoring group (PA/N) (Experimental)
  Interventions: Behavioral: Physical Activity; Behavioral: Nutrition Counseling
- Physical activity, tele-resistance training, nutrition counseling and monitoring group (RT/N) (Experimental)
  Interventions: Behavioral: Physical Activity; Behavioral: Nutrition Counseling; Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Physical Activity — Each participant will receive a Fitbit device with instruction and encouragement to self-monitor physical activity using step counts.
Behavioral: Nutrition Counseling — Participants will receive nutritional counseling with a registered dietician.
Behavioral: Resistance Training — Participants will engage in progressive, full-body resistance training based on American College of Sports Medicine (ACSM) guidelines.
  Arms: Physical activity, tele-resistance training, nutrition counseling and monitoring group (RT/N)

SUMMARY:
The purpose of the study is to examine the feasibility and acceptability of an exercise and nutrition "prehabilitation" program for patients preparing for pancreatic cancer resection (removal).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Biopsy-proven pancreatic ductal adenocarcinoma (PDAC), borderline resectable at diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Undergoing neoadjuvant chemotherapy with treatment plan including chemoradiation therapy and surgical resection
* Ability to read and speak English

Exclusion Criteria:

* Regular engagement in RT (2x/week targeting all major muscle groups)
* Screen failure for exercise safety based on PAR-Q
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease
* Recent fracture or acute musculoskeletal injury that precludes ability to participate in RT
* Numeric pain rating scale greater than or equal to a 7 out of 10
* Myopathic or rheumatologic disease that impacts physical function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of PA/N and RT/N programs | Up to 16 weeks
  The number of participants who complete T1 and T0 measures.

SECONDARY OUTCOMES:
Examine exploratory outcomes and clinical characteristics | Up to 16 weeks
  The number of participants who demonstrate improvements in exploratory outcome measures.
Compare clinical and treatment outcomes | Up to 16 weeks
  Chi-Square testing will be used to determine if there's a significant difference in outcomes between the treatment group and a usual care comparison group.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Parker, PhD, Principal Investigator — Moffitt Cancer Center; Pamela Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States